CLINICAL TRIAL: NCT03653403
Title: A Phase 1b Open-Label, Randomized Study Evaluating the Absorption and Systemic Pharmacokinetics of Topically Applied IDP-126 Gel in Comparison With Control Gel in Subjects With Acne Vulgaris Under Maximal Use Conditions
Brief Title: Open-Label, Randomized Study Evaluating the Absorption and Systemic Pharmacokinetics of Topically Applied IDP-126 Gel in Comparison With Control Gel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: V01-126A-501
Record Dates: First submitted 2018-08-20; First posted 2018-08-31 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Approximately 48 subjects who meet the study criteria will be enrolled and will receive treatment with one of the 2 study drugs. Approximately 20 subjects will be enrolled in the Control Gel treatment arm and approximately 28 subjects in the IDP-126 Gel treatment arm will be enrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- IDP-126 Gel (Experimental): Component A
  Interventions: Drug: IDP-126 Gel
- Control Gel (Active Comparator): Gel
  Interventions: Drug: Control Gel

INTERVENTIONS:
Drug: IDP-126 Gel — Component A
  Arms: IDP-126 Gel
Drug: Control Gel — gel
  Arms: Control Gel

SUMMARY:
This will be an open-label study designed to assess the safety and plasma PK of topically applied IDP-126 Gel compared to Control Gel.

DETAILED DESCRIPTION:
To evaluate the safety and plasma pharmacokinetics (PK) of clindamycin and adapalene in IDP-126 Gel compared with that from Control Gel in subjects with moderate to severe acne vulgaris (acne) during once daily topical application of IDP-126 Gel for 28 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 9 years of age (at least 12 years of age for Control Gel);
2. Verbal and signed written informed consent must be obtained. Subjects less than age of consent must sign an assent for the study and a parent or a legal guardian must sign the informed consent (if subject reaches age of consent during the study they should be re-consented at the next study visit);
3. Subject must have a score of 3 (moderate) or 4 (severe) on the Evaluator's Global Severity assessment at the screening and baseline visit

Exclusion Criteria:

1. Use of an investigational drug or device within 30 days of enrollment or participation in a research study concurrent with this study;
2. Any dermatological conditions on the face that could interfere with clinical evaluations such as acne conglobata, acne fulminans, secondary acne, perioral dermatitis, clinically significant rosacea, gramnegative folliculitis, dermatitis, eczema;
3. Any underlying disease(s) or some other dermatological condition of the face that requires the use of interfering topical or systemic therapy or makes evaluations and lesion count inconclusive;
4. Subjects with a facial beard or mustache that could interfere with the study assessments;
5. Subjects with more than two (2) facial nodules;
6. Evidence or history of cosmetic-related acne

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-06-19 (Actual); Study Completion 2019-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | All AEs will be followed from onset of the adverse event through the end of Study Day 28 visit
  During the study, subjects will be assessed for the occurrence of new and ongoing AEs. Descriptions of AEs will include the dates of onset and resolution, maximum severity, seriousness, action taken regarding study drug, corrective treatment, outcome, and investigator's assessment of causality. Worsening of disease will not be considered an AE unless it results in discontinuation of the subject from the study or requires medical intervention prohibited by the protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Anya Loncaric, Study Director — Bausch Health Companies
Locations (1):
- Valeant Site 01, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided